CLINICAL TRIAL: NCT04584450
Title: Investigation of Validity and Reliability of Post-COVID-19 Functional Status Scale
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Assoc. Prof., Hacettepe University
Other Study IDs: GO 20/788
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: COVID-19 survivors.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — data collection using questionnaire

SUMMARY:
The new type of Coronavirus (SARS-CoV-2) epidemic puts great pressure on health systems around the world. A large number of people are hospitalized in intensive care units due to acute respiratory distress syndrome due to SARS-CoV-2. Common symptoms seen with SARS-CoV-2 include fever, cough, and dyspnea, as well as pneumonia, severe acute respiratory distress syndrome, renal failure, and even death. Many patients develop mild to moderate disease without pneumonia. The respiratory condition of some patients continues to worsen gradually and develop acute respiratory distress syndrome, which usually requires mechanical ventilation support.

Exercise capacity and health status of individuals who survived severe acute respiratory distress syndrome are lower than the general population. Persistent physical, cognitive, and psychosocial disorders can be seen in people who have survived acute respiratory distress syndrome.

Given the clinical and radiological heterogeneity of COVID-19, it is important to have a simple tool for the disease to monitor the course of symptoms and the impact of symptoms on patients' functional status.

Klok FA et al. developed the Post-COVID-19 Functional Status Scale (PCFS). PCFS can be evaluated for functional sequelae after discharge from the hospital, at 4 and 8 weeks after discharge, to directly monitor recovery, and at 6 months. The aim of this study is to investigate the validity and reliability of PCFS in Turkish population. Research permission to investigate the validity and reliability of PCFS in the Turkish population was obtained from the developer of the PCFS.

ELIGIBILITY:
Inclusion Criteria:

* clinically stable,
* being 18 years of age or older,
* having education level at least primary school,
* whose local language is Turkish,
* being discharged after COVID-19
* giving consent on a voluntary basis.

Exclusion Criteria:

* having an unstable clinical condition,
* being stayed in intensive care,
* having severe neuromuscular and musculoskeletal problems,
* not being able to cooperate to fill questionnaires,
* having a cognitive problem,
* not being able to read,
* not being willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID-19 survivors
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Post-COVID-19 Functional Status Scale (Turkish version) | Through study completion, an average of 1 year
  It has been proposed as a tool to measure the full spectrum of functional outcomes following COVID-19. Post-COVID-19 Functional Status scale was reported to be used to monitor functional status. Scoring varies between 0-4. The expression 0 in PCFS indicates that there is no functional limitation. Grade 4 describes patients with severe functional limitations that require assistance with activities of daily living.

SECONDARY OUTCOMES:
Dyspnea assessment | Through study completion, an average of 1 year
  Dyspnea will be assessed by the Modified Medical Research Council (MMRC) dyspnea scale. Individuals are asked to choose the expression that best describes their dyspnea level. Scoring in MMRC varies between 0-4 points. "0 points" means that there is no dyspnea; "4 points" indicates that there is a perception of dyspnea during basic daily life activities such as dressing.
Evaluation of daily living activities | Through study completion, an average of 1 year
  The Barthel index was developed by Mahoney and Barthel in 1965. It is an index that is simple, understandable and includes all parameters of daily life activities. Its Turkish validity and reliability were made by Küçükdeveci et al. It consists of 10 sub-headings: eating, bathing, self-care, dressing, bladder control, bowel control, toilet use, chair / bed transfer, mobility, and use of stairs. Its scoring ranges from 0 to 100.
Assessment of the structural validity of the Post-COVID-19 Functional Status Scale | Through study completion, an average of 1 year
  The London Chest Activities of Daily Living Scale, developed by Garrod et al., will be used to evaluate the structural validity of the Post-COVID-19 Functional Status Scale. This questionnaire consists of 15 items and four components: personal care (4 items), housework (6 items), physical (2 items) and leisure (3 items). Each item is scored between 0 and 5. High scores show that the limitation in daily living activities is greater. The total score can reach 75 at most. The validity and reliability study of the questionnaire for the Turkish population has been conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, Study Chair — Hacettepe University; Gülay Sain-Güven, Study Chair — Hacettepe University; Naciye Vardar-Yagli, Study Chair — Hacettepe University; Melda Saglam, Study Chair — Hacettepe University; Lale Özışık, Study Chair — Hacettepe University; Nursel Çalık-Başaran, Study Chair — Hacettepe University; Oğuz Abdullah Uyaroğlu, Study Chair — Hacettepe University; Aslıhan Çakmak, Principal Investigator — Hacettepe Üniversitesi; Esra Kınacı, Principal Investigator — Hacettepe University; Ebru Çalık-Kütükcü, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306